CLINICAL TRIAL: NCT05260216
Title: Clinical Analysis of Cariogram and Cariostat for Risk Assessment and Comprehensive Intervention of Early-childhood-caries
Brief Title: Clinical Analysis of a Risk-graded and Comprehensive Intervention for Early-childhood-caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CARGACIFECC
Record Dates: First submitted 2021-12-12; First posted 2022-03-02 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-12

CONDITIONS: Early Childhood Caries
Keywords: Caries risk assessment
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After the data is entered, the analyst is analyzed under the premise of uninformed, and the packet is performed after all analyzes are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental subgroup of Cariostat (Experimental): Use Cariostat as the caries risk assessment tool to divide the children into different risk levels. Based on the results, children with low risk of caries will receive twice fluoride foam each year and oral hygiene guidance, children with middle or high risk of caries will receive forth fluoride applications each year, oral hygiene guidance and professional caries treatment.
  Interventions: Combination Product: Comprehensive prevention and treatment
- Experimental subgroup of Cariogram (Experimental): Use Cariogram as the caries risk assessment tool to divide the children into different risk levels. Based on the results, children with low risk of caries will receive twice fluoride foam each year and oral hygiene guidance, children with middle or high risk of caries will receive forth fluoride applications each year, oral hygiene guidance and professional caries treatment.
  Interventions: Combination Product: Comprehensive prevention and treatment
- Control group (Placebo Comparator): Use Cariogram and as the caries risk assessment tool to divide the children into different risk levels. All children will receive routine prevention including wice fluoride foam each year and oral hygiene guidance.
  Interventions: Combination Product: Routine prevention

INTERVENTIONS:
Combination Product: Comprehensive prevention and treatment — Children with low risk of caries will receive routine prevention including fluoride foam application twice a year and oral hygiene guidance. Children with middle or high risk of caries will receive fluoride varnish application twice a year and caries restorative treatment in addition to routine prevention. The risk-graded intervention is one kind of comprehensive prevention and treatment.
  Arms: Experimental subgroup of Cariogram; Experimental subgroup of Cariostat
Combination Product: Routine prevention — Routine prevention includes fluoride foam application twice a year and oral hygiene guidance.
  Arms: Control group

SUMMARY:
Cariogram and Cariostat will be used to assess the risk of caries in kindergarten children aged 3 years. Routine preventive measures will be taken for children at low risk of caries, and intensive intervention measures will be taken for children at medium and high risk. Routine measures will be taken for the control group. After one and two year, the prevalence of caries in the experimental group and the control group should be evaluated, and the cost-effectiveness evaluation will be conducted.

DETAILED DESCRIPTION:
Caries risk-graded intervention for preschool children is needed as different child has different risk to suffer from caries.

Cariogram and Cariostat are two different and common caries risk assessment tools. Cariogram is a complicated but economical computer program which is more sensitive for caries risk assessment. Cariostat is a biological reagents with high specificity but it may be expensive to use for large numbers of children.

The experimental group will be divided into two subgroups, one use Cariogram and the other use Cariostat to assess the risk. Based on the results of the assessment, children with low risk of caries will get routine prevention including twice fluorinated foams each year and hygiene. Children with middle or high risk of caries will receive twice fluorinated varnish each year and professional caries treatment in addition to routine prevention.Routine prevention will be taken for the control group with both Cariogram and Cariostat assessment.

Follow-up will arrange one and two years after baseline recruitment. All participants will receive oral health-related questionnaires at baseline and follow-up.

The prevalence of caries in the experimental group and the control group should be evaluated, and the cost-effectiveness evaluation will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Junior kindergarten children who enter the kindergarten in September 2021 and can cooperate with the oral health examination.
2. Parents of children fully understand the purpose of the study, cooperate with the questionnaire survey during the study, give informed consent and sign the informed consent form.
3. The child has no serious systemic diseases, has not taken hormones and immunosuppressants within 6 months, and has no history of antibiotic use within 1 month，and is not allergic to fluoride.

Exclusion Criteria:

1. Parents of children refuse to provide information about children's oral health or questionnaires.
2. Children cannot cooperate with oral health examination.
3. The child has a serious systemic disease that may affect the results of the study.
4. Children who are allergic to fluoride.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Decay teeth,Missed teeth and filled teeth (DMFT) and the change between different time points. | Baseline, one year follow up and two year follow up.
  The average value of the sum of the number of decayed teeth, the number of filled teeth, and the number of missed teeth due to caries.

SECONDARY OUTCOMES:
Caries prevalence and the change between different time points. | Baseline, one year follow up and two year follow up.
  The proportion of population with caries in the whole participants.

CONTACTS AND LOCATIONS:
Overall Officials: Menglin Cheng, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, informed consent form and clinical study report are to be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When the two years follow up is completed and the result and conclusion of the study is published, the data will become available for half a year.
Access Criteria: The sharing criteria in this study is to the research leader who register study with key words of Caries Risk Assessment on the Clinical Trail.